CLINICAL TRIAL: NCT02291549
Title: A Clinical Evaluation of the Safety and Efficacy of the Steroid-Releasing S8 Sinus Implant in Chronic Sinusitis Patients With Recurrent Sinus Obstruction
Brief Title: S8 Sinus Implant in Chronic Sinusitis Patients With Recurrent Nasal Polyps
Acronym: RESOLVE_II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P500-1113
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Chronic Sinusitis; Nasal Polyposis
Keywords: endoscopic sinus surgery; corticosteroid; chronic rhinosinusitis; mometasone furoate; polyposis
MeSH Terms: conditions — Nasal Polyps | interventions — Mometasone Furoate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blindfolded and earmuffed during the baseline procedure and follow-up endoscopic examinations. Implants were removed at Day 60 to allow blinded assessment of bilateral polyp grade at Day 90 by a centralized videoendoscopy review by a panel of 3 independent sinus surgeons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Mometasone furoate nasal spray (200mcg) once daily
  Interventions: Drug: S8 Sinus Implant; Drug: Mometasone furoate nasal spray
- Control (Sham Comparator): In-office bilateral sham procedure
  Mometasone furoate nasal spray (200mcg) once daily
  Interventions: Drug: Mometasone furoate nasal spray; Procedure: Sham

INTERVENTIONS:
Drug: S8 Sinus Implant — In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Other Names: SINUVA (mometasone furoate) sinus implant
  Arms: Treatment
Drug: Mometasone furoate nasal spray — Mometasone furoate nasal spray (200mcg) once daily
  Other Names: Nasonex
Procedure: Sham — In-office bilateral sham procedure, consisting of advancement of a delivery system with the S8 Sinus Implant into the ethmoid sinuses followed by removal without deployment.
  Other Names: Sham procedure
  Arms: Control

SUMMARY:
The RESOLVE II Study is a randomized, single-blind, parallel arm, concurrently controlled, multicenter study with 300 chronic sinusitis patients who had prior endoscopic sinus surgery but present with recurrent sinus obstruction.

DETAILED DESCRIPTION:
The RESOLVE II Study is a randomized, sham-controlled, double-blind, parallel arm multicenter trial conducted in up to 45 clinical centers (academic and private) across the United States in 300 adults with chronic sinusitis, who are indicated for revision surgery because of recurring nasal obstruction/congestion symptoms and bilateral ethmoid polyposis.

ELIGIBILITY:
Key inclusion criteria:

* Confirmed diagnosis of chronic sinusitis
* Patient has undergone bilateral total ethmoidectomy at least 90 days prior to screening
* Patient has Nasal Obstruction/Congestion score of at least 2 (scale from 0 to 3) on at least 5 days during the 7 days following informed consent, despite use of topical intranasal steroid irrigations or sprays for at least 14 days preceding scoring, as documented in medication records
* Indication for repeat ESS:

  * Complaints of at least 2 symptoms of chronic sinusitis: nasal obstruction/congestion, post-nasal discharge, thick nasal discharge, facial pain/pressure, or decreased sense of smell
  * Endoscopic evidence of bilateral sinus obstruction due to polyposis (minimum grade 2 on each side)
  * History of high-dose steroid use and/or sinus steroid irrigations within the preceding 1 year

Exclusion criteria:

* Patient has presence of polyposis grade 1, 1.5 or 4 on either side
* Patient has presence of adhesions/synechiae grades 3 or 4
* Patient has known history of immune deficiency
* Patient has concurrent condition such as cancer or HIV requiring active chemotherapy and/or immunotherapy management for the disease
* Patient has oral-steroid dependent condition such as COPD, asthma or other condition
* Patient has known history of allergy or intolerance to corticosteroids or mometasone furoate
* Patient has presence of physical obstruction that would preclude access to either ethmoid sinus for implant delivery (e.g., severe septal deviation, septal spur, very small middle meatus, total obstruction of the nasal passage with severe scarring, polyposis)
* Patient has clinical evidence of acute bacterial sinusitis
* Patient has clinical evidence or suspicion of invasive fungal sinusitis
* Patient has evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 90-day follow-up period
* Patient is currently participating in another clinical trial or has already participated in this clinical trial
* Patient has history of insulin dependent diabetes mellitus
* Patient has previously undergone ESS and experienced a cerebrospinal fluid (CSF) leak or has residual compromised vision as a result of a complication in a prior ESS procedure
* Patient has known dehiscence of the lamina papyracea
* Patient has evidence of active viral illness
* Patient has known history or diagnosis of glaucoma or ocular hypertension (prior ocular exam with IOP>21 mm Hg and pressure lowering medication given) or posterior subcapsular cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Kern, MD, Principal Investigator — Department of Otolaryngology, Northwestern University, Chicago, IL; Jose P. Stolovitzky, MD, Principal Investigator — ENT of Georgia, Atlanta, GA
Locations (40):
- United States (40):
  - The University of Alabama Birmingham, Birmingham, Alabama
  - Kaiser Permanente Orange County Irvine Medical Center, Irvine, California
  - Sacramento Ear, Nose and Throat Surgical and Medical Group, Inc., Sacramento, California
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - GW Medical Facility Associates, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - South Florida ENT, Miami, Florida
  - & Facial Plastic Surgery, Riverview, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Northwestern Medical Faculty Foundation, Department of Otolaryngology, Chicago, Illinois
  - DuPage Medical Group, Naperville, Illinois
  - Iowa ENT Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Associated Surgical Specialists, Covington, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - Rontal Akervall Clinic, Royal Oak, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ear, Nose and Throat Consultants of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Breathe America/NM Sinus, Albuquerque, New Mexico
  - Albany ENT & Allergy, Albany, New York
  - Madison ENT & Facial Plastic Surgery, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Charlotte Eye, Ear, Nose and Throat Associates, Concord, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Bethlehem Ear, Nose and Throat Associates, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, Houston, Texas
  - Cache Valley ENT, North Logan, Utah
  - Intermountain/ENT Center of UT, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Reston ENT, Reston, Virginia
  - Virginia ENT, Richmond, Virginia
  - Medical College of Wisconsin - Greenway Clinic, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kern RC, Stolovitzky JP, Silvers SL, Singh A, Lee JT, Yen DM, Iloreta AMC Jr, Langford FPJ, Karanfilov B, Matheny KE, Stambaugh JW, Gawlicka AK; RESOLVE II study investigators. A phase 3 trial of mometasone furoate sinus implants for chronic sinusitis with recurrent nasal polyps. Int Forum Allergy Rhinol. 2018 Apr;8(4):471-481. doi: 10.1002/alr.22084. Epub 2018 Jan 19. PMID 29350840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 40 sites across the US between December 2014 and May 2016, of which 34 sites enrolled at least 1 patient.
Pre-assignment Details: Patients were considered enrolled into the study after signing the ICF and entered a 2-week screening period. A video-recorded screening endoscopy and symptom scoring, using a daily diary, were required to confirm patient eligibility. Video-endoscopies were assessed by an independent reviewer in order to confirm bilateral polyposis.
Groups:
- S8 Sinus Implant: Bilateral in-office placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Mometasone furoate nasal spray (200 mcg) once daily
- Control: Bilateral in-office sham procedure
  Mometasone furoate nasal spray (200 mcg) once daily
Period: Overall Study
Arm/Group | S8 Sinus Implant | Control
Started | 201 | 99
Completed | 200 | 98
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 201 | 99 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (12.9) | 47.9 (12.4) | 49.6 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 43 | 117
  Male | 127 | 56 | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 164 | 80 | 244
  Race/Ethnicity: Black | 27 | 13 | 40
  Race/Ethnicity: Asian | 4 | 4 | 8
  Race/Ethnicity: Other | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Nasal Obstruction/Congestion Score
Description: Determined by patients using a daily diary on a scale from 0 (no symptoms) to 3 (severe symptoms) over a period of 7 days prior to the baseline and Day 30 visits. Negative values for change from baseline indicate reduction (improvement) in nasal obstruction/congestion symptoms.
Time Frame: Day 30
Population: Intent-to-treat population. Scoring for >=4 days in 7 days before the baseline and Day 30 visits was required. Sensitivity analyses, including tipping point, were prespecified if missing values exceed 5%. There were 4 (1.3%) participants (2 treatment, 2 control) with missing values at Day 30. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
units on a scale
  Baseline: number analyzed (Participants) | 200 | 99
  Baseline | 2.36 (0.488) | 2.35 (0.479)
  30 Day: number analyzed (Participants) | 199 | 97
  30 Day | 1.56 (0.743) | 1.79 (0.674)
  Change from baseline: number analyzed (Participants) | 199 | 97
  Change from baseline | -0.80 (0.729) | -0.56 (0.619)
Statistical Analysis 1: Comparison: Treatment vs Control; ANCOVA model with site and treatment group as fixed effects and contrasts constructed to estimate the difference between treatment groups. The primary efficacy hypothesis was that the use of the S8 Sinus Implant would reduce the Nasal Obstruction/Congestion score compared to the control group. The null hypothesis was H0: β1=0 and alternative hypothesis was H1: β1 ≠ 0. Only a statistically significant, negative estimate of β1 was to constitute evidence of effectiveness; Test type: Superiority; p = 0.0074, ANCOVA — The 2-sided alpha was 0.05. P-value was not adjusted for multiple comparison; Where appropriate, confidence intervals of the difference were constructed using the estimate of the least-squares means; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.39 to -0.06]

2. Primary Outcome: Bilateral Polyp Grade
Description: Polyp grade was determined by an independent panel of 3 sinus surgeons based on a centralized, blinded videoendoscopy review. Each sinus was graded from 0 (no visible polyps) to 4 (nasal polyps completely obstructing nasal cavity) and then the left and right values were added to obtain a total bilateral polyp grade, ranging from 0 to 8. Negative values for change from baseline indicated reduction (improvement) in bilateral polyp grade.
Time Frame: Day 90
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. Sensitivity analyses, including tipping point, were prespecified if missing values exceed 5%. There were 8 (2.7%) participants (6 treatment, 2 control) with missing values at Day 90. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment: In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Mometasone furoate nasal spray (200 mcg) once daily
- Control: In-office bilateral sham procedure
  Mometasone furoate nasal spray (200 mcg) once daily
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
units on a scale
  Baseline | 5.48 (1.132) | 5.43 (1.009)
  Day 90: number analyzed (Participants) | 195 | 97
  Day 90 | 4.91 (1.432) | 5.26 (1.378)
  Change from baseline: number analyzed (Participants) | 195 | 97
  Change from baseline | -0.56 (1.059) | -0.15 (0.907)
Statistical Analysis 1: Comparison: Treatment vs Control; The between treatment group difference was estimated using the ANCOVA model with site and treatment group as fixed effects. The primary efficacy hypothesis was that the use of the S8 Sinus Implant would reduce the bilateral polyp grade compared to the control group. The null hypothesis was H0: β1=0 and alternative hypothesis was H1: β1 ≠ 0. Only a statistically significant, negative estimate of β1 was to constitute evidence of effectiveness; Test type: Superiority; p = 0.0073, ANCOVA — The 2-sided alpha was 0.05. P-value was not adjusted for multiple comparisons; ANCOVA model with site and treatment group as fixed effects and contrasts constructed to estimate the difference between treatment groups; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.60 to -0.09]

3. Secondary Outcome: Percentage of Patients Indicated for Repeat Endoscopic Sinus Surgery (RESS)
Description: Proportion of patients still indicated for RESS at day 90 despite ongoing use of mometasone furoate nasal spray based on clinical investigator assessment using study-specific criteria. To be indicated for RESS, patients had to: (1) complain of nasal obstruction/congestion (moderate to severe) and postnasal discharge, facial pain/pressure/fullness, or altered sense of smell/taste; (2) have endoscopic evidence of persisting nasal polyps (grade >= 2 on each side); and (3) have received (required at baseline) or need a systemic steroid as noted during endoscopy.
Time Frame: Day 90
Population: Intent-to-treat population, consisting of all patients in whom an implant or sham procedure was attempted. 2 participants did not complete Day 90 visit. No imputation of missing values was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
Participants
  Baseline | 201 | 99
  Day 90: number analyzed (Participants) | 200 | 98
  Day 90 | 78 | 62
Statistical Analysis 1: Comparison: Treatment vs Control; Test: H0: OR = 1 vs. OR ≠ 1 by Cochrane-Mantel-Haenszel test; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — P-value adjusted for multiplicity using the Holm's step-down procedure at a 2-sided significance level of 0.05; Adjusted p-value is presented; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.63 to 4.44]

4. Secondary Outcome: Ethmoid Sinus Obstruction
Description: Percentage of the ethmoid sinus volume obstructed by scarring, polyps, or edema on endoscopy, as determined by an independent panel of 3 sinus surgeons based on a centralized, blinded videoendoscopy review using a 100-mm visual analogue scale (VAS), ranging from 0 (absence of obstruction) to 100 (complete obstruction). Negative values for change from baseline indicated reduction (improvement) in ethmoid sinus obstruction.
Time Frame: Day 90
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 8 (2.7%) participants (6 treatment, 2 control) with missing values at Day 90. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
units on a scale
  Baseline | 69.2 (19.87) | 67.0 (18.55)
  Day 90: number analyzed (Participants) | 195 | 97
  Day 90 | 57.7 (23.57) | 64.8 (23.14)
  Change from baseline | -11.3 (18.11) | -1.9 (14.36)
Statistical Analysis 1: Comparison: Treatment vs Control; ANCOVA model with site and treatment group as fixed effects and contrasts constructed to estimate the difference between treatment groups.The null hypothesis was H0: β1 = 0 and the alternative hypothesis was H1: β1 ≠ 0. Although the alternative hypothesis was specified as 2-sided, only a statistically significant, negative estimate of β1 constituted evidence of effectiveness. The 2-sided alpha for this test was 0.05; Test type: Superiority; p = 0.0007, ANCOVA — P-value adjusted for multiplicity using the Holm's step-down procedure at a 2-sided significance level of 0.05; Adjusted p-value is presented; Mean Difference (Final Values) = -7.96, 95% CI 2-sided [-12.10 to -3.83]

5. Secondary Outcome: Nasal Obstruction/Congestion Score
Description: Determined by patients using a daily diary on a scale from 0 (no symptoms) to 3 (severe symptoms) over a period of 7 days prior to baseline and Day 90. Negative values for change from baseline indicated reduction (improvement) in nasal obstruction/congestion symptoms.
Time Frame: Day 90
Population: Intent-to-treat population. Scoring for >=4 of 7 days immediately preceding the baseline and Day 90 visits was required. There were 34 (11.3%) participants with missing scores: 23 treatment and 10 control at Day 90 and 1 (treatment) at baseline. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
units on a scale
  Baseline: number analyzed (Participants) | 200 | 99
  Baseline | 2.36 (0.488) | 2.35 (0.479)
  Day 90: number analyzed (Participants) | 178 | 89
  Day 90 | 1.42 (0.814) | 1.68 (0.812)
  Change from baseline: number analyzed (Participants) | 177 | 89
  Change from baseline | -0.93 (0.798) | -0.69 (0.791)
Statistical Analysis 1: Comparison: Treatment vs Control; ANCOVA model with site and treatment group as fixed effects and contrasts constructed to estimate the difference between treatment groups. The null hypothesis was H0: β1=0 and the alternative hypothesis was H1: β1 ≠ 0. Only a statistically significant, negative estimate of β1 was to constitute evidence of effectiveness; Test type: Superiority; p = 0.0248, ANCOVA — P-value adjusted for multiplicity using the Holm's step-down procedure at a 2-sided significance level of 0.05; Adjusted p-value is presented; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.48 to -0.07]

6. Secondary Outcome: Decreased Sense of Smell Score
Description: Determined by patients on a 6-point Likert scale from 0 (absent) to 5 (very severe). Negative values for change from baseline indicated reduction (improvement) in sense of smell.
Time Frame: Day 90
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 5 (1.7%) participants (3 treatment, 2 control) with missing values at Day 90. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
units on a scale
  Baseline | 4.1 (1.38) | 4.1 (1.36)
  Day 90: number analyzed (Participants) | 198 | 97
  Day 90 | 2.9 (1.96) | 3.4 (1.86)
  Change from baseline: number analyzed (Participants) | 198 | 97
  Change from baseline | -1.20 (1.659) | -0.76 (1.599)
Statistical Analysis 1: Comparison: Treatment vs Control; ANCOVA model with site and treatment group as fixed effects and contrasts constructed to estimate the difference between treatment groups. The null hypothesis was H0: β1=0 and alternative hypothesis was H1: β1 ≠ 0. Only a statistically significant, negative estimate of β1 was to constitute evidence of effectiveness; Test type: Superiority; p = 0.0470, ANCOVA — P-value adjusted for multiplicity using the Holm's step-down procedure at a 2-sided significance level of 0.05; The adjusted p-value is presentenced; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.85 to -0.06]

7. Secondary Outcome: Facial Pain/Pressure Score
Description: Determined by patients on a 6-point Likert scale from 0 (absent) to 5 (very severe). Negative values for change from baseline indicated reduction (improvement) in facial pain/pressure symptoms.
Time Frame: Day 90
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 5 (1.7%) participants (3 treatment, 2 control) with missing values: 3 at baseline (1 treatment, 1 control)) and 2 at Day 90 (1 treatment, 1 control) No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 201 | 99
units on a scale
  Baseline: number analyzed (Participants) | 200 | 98
  Baseline | 1.9 (1.40) | 2.2 (1.42)
  Day 90: number analyzed (Participants) | 198 | 97
  Day 90 | 1.1 (1.25) | 1.2 (1.20)
  Change from baseline: number analyzed (Participants) | 197 | 96
  Change from baseline | -0.77 (1.209) | -0.90 (1.269)
Statistical Analysis 1: Comparison: Treatment vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.9130, ANCOVA — P-value adjusted for multiplicity using the Holm's step-down procedure at a 2-sided significance level of 0.05; Adjusted p-value is presented

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/99
Serious Adverse Events (participants affected / at risk) | 1/201 | 0/99
Other Adverse Events (participants affected / at risk) | 53/201 | 28/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=201) | Control (N=99)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — SAE that was judged to be related to the S8 Sinus Implant
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=201) | Control (N=99)
Acute Sinusitis (Infections and infestations) | 22 | 12
Chronic Sinusitis (Infections and infestations) | 10 | 8
Upper respiratory tract infection (Infections and infestations) | 11 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 4

LIMITATIONS AND CAVEATS:
1. The absence of a defined medical regimen prior to enrollment.
2. The clinical investigators performing assessment of indication for RESS at Day 90 were unblinded.
3. The relatively short duration of the trial (90 days).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No